CLINICAL TRIAL: NCT04027075
Title: Mindfulness Mobile App to Reduce Adolescent Substance Use
Acronym: Qlarity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA043288-02
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Drinking; Adolescent Problem Behavior
Keywords: Adolescent; Alcohol; Marijuana; Mindfulness
MeSH Terms: conditions — Underage Drinking; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: This study will recruit 400 adolescents to test an app designed to increase mindfulness skills and reduce substance use. Participants will be randomly assigned in equal numbers to the intervention group (and will use the app) or the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will be asked to use the Qlarity app daily in the month following the baseline assessment. This group will also receive services as usual from the Department of Youth Services.
  Interventions: Behavioral: Qlarity app users
- Services as usual (No Intervention): This group will receive services as usual from the Department of Youth Services.

INTERVENTIONS:
Behavioral: Qlarity app users — Use of the Qlarity app involves completing 12 modules and 12 practice sessions over 30 days.
  Arms: Intervention

SUMMARY:
Substance-abusing youth - especially those who are involved in the juvenile justice system - are at higher risk than nonusers for mental health problems, including depression, conduct problems, personality disorders, suicidal thoughts, attempted suicide, and completed suicide. The proposed Phase II project aims to develop and test the efficacy of a mobile app, called Qlarity, that is geared toward helping high risk adolescent substance users reduce or quit their substance use. The Qlarity app is based on the primary substance use cessation components tested in our previous work with juvenile justice-involved adolescents and on intervention components shown to be central to smoking cessation; it applies a mindfulness approach as the guiding framework for the intervention.

DETAILED DESCRIPTION:
There is growing evidence that interventions based on mindfulness have been an efficacious intervention for a variety of problems, including substance use among adolescents. We propose to adapt and test the feasibility and efficacy of a smart phone application (app) intervention prototype that would help adolescent substance users reduce or quit their substance use through the development of stress reduction, emotion regulation, and mindfulness skills. During the development process, 20 high-risk adolescents will be recruited for participation in focus groups and usability testing of early versions of the app; their initial reactions to content and functionality will help guide final iterations. Qlarity is a twelve module program, and each module consists of a teaching component and a practice component. Modules take 5 minutes or less to complete. Module topics include developing an awareness of mind and body states, mindful decision making, and maintaining sobriety.

In this study, the Qlarity app will be evaluated with 400 high risk adolescents that are involved in the juvenile justice system; the first 20 adolescents will be involved in the development process and the remaining 380 participants will be randomly and equally assigned to the Qlarity condition (n = 190) or the Department of Youth Services standard treatment condition (n = 190). Youth will be assessed at baseline and will be instructed to attempt to reduce substance use with a target quit date of 28 days in the future. The Qlarity group will receive instructions for using the app in the 28 days following baseline. All youth will complete 1 and 3 month follow-ups. Assessments will consist of online surveys asking about substance use, emotion regulation, family demographics, and mindfulness practices. The Qlarity group will also be asked for their thoughts and opinions on the app. Biochemical verification of self-reported substance use, a urine sample, will be collected at each interview.

ELIGIBILITY:
Inclusion Criteria:

* any gender, age 13-18
* recent involvement with juvenile justice system
* documented substance use
* English speaking
* living in the community (e.g., with biological/adoptive/foster parents)

Exclusion Criteria:

* non-English speaking

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 257 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Smith, PhD, Principal Investigator — Oregon Research Behavioral Intervention Strategies
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Springfield, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Services as Usual
Started | 129 | 128
Completed | 88 | 106
Not Completed | 41 | 22
Not completed — Lost to Follow-up | 41 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Services as Usual | Total
Number analyzed (Participants) | 129 | 128 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.30 (1.62) | 15.23 (1.68) | 15.26 (1.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 101
  Male | 79 | 77 | 156
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 9 | 14 | 23
  White | 96 | 81 | 177
  More than one race | 12 | 14 | 26
  Unknown or Not Reported | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Marijuana Use
Description: An EZ Split Key 10 panel cup was used to detect marijuana in a urine sample.
Time Frame: Baseline, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
Participants
  Baseline | 47 | 40
  3 months | 41 | 41
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .962, Chi-squared; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.51 to 2.02] — The odds ratio applies to the group comparison (Intervention vs. Services as Usual) at 3-months. Group was coded 1 = Intervention and 0 = Services as Usual

2. Primary Outcome: Number of Participants With Prescribed Drugs Use
Description: An EZ Split Key 10 panel cup was used to detect prescribed drugs in a urine sample.
Time Frame: Baseline, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
Participants
  Baseline | 55 | 46
  3 months | 22 | 27
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .109, Chi-squared; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.19 to 1.18] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Number of Participants With Hard Drug Use
Description: An EZ Split Key 10 panel cup was used to detect hard drugs in a urine sample.
Time Frame: Baseline, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
Participants
  Baseline | 22 | 14
  3 months | 15 | 14
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .227, Chi-squared; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.75 to 3.29] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Change in Adolescent Use of Cigarettes
Description: Change in nicotine use (frequency of use and amount consumed) as measured by Youth Substance Use Interview
Time Frame: Baseline, 1 month, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
Participants
  Baseline | 20 | 14
  1 month | 13 | 12
  3 month | 16 | 13
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .681, Chi-squared; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.50 to 2.87] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Change in Adolescent Use of Alcohol
Description: Change in alcohol use (frequency of use and amount consumed) as measured by Youth Substance Use Interview
Time Frame: Baseline, 1 month, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
Participants
  Baseline | 23 | 15
  1 month | 10 | 12
  3 months | 18 | 17
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .650, Chi-squared; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.58 to 2.42] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Change in Adolescent Use of Marijuana
Description: Change in marijuana use (frequency of use and amount consumed) as measured by Youth Substance Use Interview
Time Frame: Baseline, 1 month, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
Participants
  Baseline | 52 | 35
  1 month | 29 | 35
  3 months | 40 | 35
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .304, Chi-squared; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.73 to 2.73] — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Change in Adolescent Use of Other Recreational Substances
Description: Change in use of hard drugs as measured by the Youth Substance Use Interview
Time Frame: Baseline, 1 month, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
Participants
  Baseline | 52 | 54
  1 month | 16 | 17
  3 months | 18 | 17
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = 0.97, Chi-squared; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.69 to 3.00] — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Change in Ability to Limit Substance Use
Description: Self-efficacy for limiting substance use consists of 6 items that assess the ability to abstain from drug use. Response options range from 0 = cannot do at all to 10 = certainly can do. A sum score was computed and thus, values can range between 0 and 60. Higher scores indicate greater ability to abstain
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
units on a scale
  Baseline | 46.60 (11.72) | 43.34 (14.23)
  1 month | 47.08 (12.63) | 47.27 (13.20)
  3 months | 44.36 (13.84) | 46.49 (12.57)
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .005, t-test, 2 sided; Mean Difference (Final Values) = -1.78, Standard Error of Mean 0.64 — The mean difference applies to the group comparison (Intervention vs. Services as Usual) in trajectory differences from baseline through 3-months. Group was coded 1 = Intervention and 0 = Services as Usual

9. Primary Outcome: Change in Emotion Regulation
Description: Emotion Regulation is measured by the Difficulties in Emotion Regulation Scale. Emotional regulation was assessed with a 5-point response option (1 = almost never, 5 = almost always). A sum score was computed and thus, values can range between 1 and 55. A higher score indicates greater levels of emotional regulation.
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
units on a scale
  Baseline | 30.93 (26.75) | 30.38 (25.88)
  1 month | 31.28 (24.71) | 34.87 (24.05)
  3 months | 28.23 (25.44) | 30.31 (25.89)
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .460, t-test, 2 sided; Mean Difference (Final Values) = -0.80, Standard Error of Mean 1.09 — [estimate comment as in outcome 8, analysis 1]

10. Primary Outcome: Change in Mindfulness Behavior - Observing Subscale
Description: Mindfulness is measured by the Five Facet Mindfulness Questionnaire. Mindfulness was assessed with a 5-point response option (1 = never or very rarely true, 5 = every often or always true) and sum scores were computed for each subscale. Subscales include observing (8 items), describing (8 items), acting with awareness (8 items), non-judging of inner experience (8 items), and non-reactivity to inner experience (7 items). Score could range from 8 to 40 for all subscales other than reactivity to inner experience which could range from 7 to 35. A higher score indicates greater levels of mindfulness.
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
units on a scale
  Baseline | 25.57 (7.55) | 25.18 (5.90)
  Pretest | 25.29 (6.15) | 24.98 (6.03)
  Posttest | 25.91 (5.74) | 25.05 (6.10)
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .851, t-test, 2 sided; Mean Difference (Final Values) = 0.05, Standard Error of Mean 0.26 — [estimate comment as in outcome 8, analysis 1]

11. Primary Outcome: Change in Mindfulness Behavior - Describing Subscale
Description: as for outcome 10
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
units on a scale
  Baseline | 24.14 (5.45) | 23.39 (5.61)
  1 month | 23.63 (6.15) | 23.26 (5.81)
  3 months | 24.22 (5.68) | 23.41 (5.67)
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .977, t-test, 2 sided; Mean Difference (Final Values) = -0.01, Standard Error of Mean 0.23 — [estimate comment as in outcome 8, analysis 1]

12. Primary Outcome: Change in Mindfulness Behavior - Acting With Awareness Subscale
Description: as for outcome 10
Time Frame: Baseline, 1 month, 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
units on a scale
  Baseline | 21.86 (5.88) | 22.16 (6.07)
  1 month | 21.93 (6.02) | 23.38 (6.16)
  3 months | 22.49 (5.73) | 22.88 (6.35)
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .456, t-test, 2 sided; Mean Difference (Final Values) = 0.20, Standard Error of Mean 0.27 — [estimate comment as in outcome 8, analysis 1]

13. Primary Outcome: Change in Mindfulness Behavior - Non-judging of Inner Experience Subscale
Description: as for outcome 10
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
units on a scale
  Baseline | 25.62 (6.98) | 25.53 (7.26)
  1 month | 26.49 (7.29) | 25.49 (7.67)
  3 months | 25.57 (7.65) | 25.55 (6.69)
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .874, t-test, 2 sided; Mean Difference (Final Values) = 0.05, Standard Error of Mean 0.31 — [estimate comment as in outcome 8, analysis 1]

14. Primary Outcome: Change in Mindfulness Behavior - Non-reactivity to Inner Experience Subscale
Description: as for outcome 10
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
units on a scale
  Baseline | 19.97 (4.60) | 19.72 (4.56)
  1 month | 20.21 (5.16) | 19.60 (4.93)
  2 month | 21.07 (4.72) | 19.59 (4.71)
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .069, t-test, 2 sided; Mean Difference (Final Values) = 0.44, Standard Error of Mean 0.24 — [estimate comment as in outcome 8, analysis 1]

15. Primary Outcome: Change in Attitude Toward Substance Use - Beliefs and Consequences Subscale
Description: Change in attitude related to drug use is measured with Adolescent Attitudes toward Substance Use. Subscales are (1) Beliefs and Consequences (9 items) and (2) Lifestyle and Value incompatibility (5 items). Response options were 0 to 10. Standardized scores were computed and values could range from -2.0 to 2.0. Higher scores represent more prosocial attitudes.
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
units on a scale
  Baseline | -0.04 (0.45) | 0.05 (0.47)
  1 month | 0.01 (0.53) | -0.01 (0.49)
  3 months | -0.00 (0.45) | 0.03 (0.52)
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .658, t-test, 2 sided; Mean Difference (Final Values) = 0.01, Standard Error of Mean 0.02 — [estimate comment as in outcome 8, analysis 1]

16. Primary Outcome: Change in Attitudes Towards Substance Use - Lifestyle and Value Incompatibility Subscale
Description: as for outcome 15
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Services as Usual
Number analyzed (Participants) | 129 | 128
units on a scale
  Baseline | -0.04 (0.57) | -0.01 (0.65)
  1 month | -0.01 (0.60) | -0.02 (0.60)
  3 months | -0.04 (0.56) | 0.03 (0.66)
Statistical Analysis 1: Comparison: Intervention vs Services as Usual; Test type: Superiority; p = .783, t-test, 2 sided; Mean Difference (Final Values) = -0.01, Standard Error of Mean 0.03 — [estimate comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the 3 month period that participants were involved in the study. Data was assessed for adverse events at all data collection timepoints: baseline, 1 month follow up, and 3 month follow up.
Arm/Group | Intervention | Services as Usual
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/128
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/128
Other Adverse Events (participants affected / at risk) | 0/129 | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT04027075/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT04027075/ICF_001.pdf